CLINICAL TRIAL: NCT00660907
Title: A 52-Week International, Multi-centre, Randomised, Parallel-group, Double-blind, Active-controlled, Phase III Study With a 156-Week Extension Period to Evaluate the Efficacy and Safety of Dapagliflozin in Combination With Metformin Compared With Sulphonylurea in Combination With Metformin in Adult Patients With Type 2 Diabetes Who Have Inadequate Glycaemic Control on Metformin Therapy Alone.
Brief Title: Efficacy and Safety of Dapagliflozin in Combination With Metformin in Type 2 Diabetes Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1690C00004
Record Dates: First submitted 2008-04-15; First posted 2008-04-17 (Estimated); Results first posted 2013-08-23 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes
Keywords: Dapagliflozin; efficacy; safety; metformin; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Glipizide; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): dapagliflozin plus metformin
  Interventions: Drug: dapagliflozin; Drug: metformin hydrochloride
- 2 (Active Comparator): glipizide plus metformin
  Interventions: Drug: glipizide; Drug: metformin hydrochloride

INTERVENTIONS:
Drug: dapagliflozin — Tablet oral 2.5, 5, or 10 mg total daily dose once daily 208 weeks
  Arms: 1
Drug: glipizide — Capsule oral 5, 10, or 20 mg total daily dose once or split/twice daily 208 weeks
  Other Names: Glucotrol
  Arms: 2
Drug: metformin hydrochloride — Tablet oral 1500, 2000, or 2500 mg total daily dose split/twice daily 218 weeks
  Other Names: Glucophage

SUMMARY:
This study is being carried out to see if dapagliflozin as an addition to metformin is effective and safe in treating patients with type 2 diabetes when compared to glipizide (sulphonylurea) as an addition to metformin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes
* Treated with oral anti-diabetic drug therapy therapy including Metformin for at least 8 weeks prior to enrolment
* HbA1c >6.5% and </=10%

Exclusion Criteria:

* Type 1 Diabetes
* Insulin therapy within one year of enrolment
* Renal (kidney) failure or dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1217 (Actual)
Dates: Start 2008-03; Primary Completion 2009-12 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Nauck, Prof. Dr. med., Principal Investigator — Diabeteszentrum Bad Lauterberg, Germany
Locations (76):
- Argentina (9):
  - Research Site, Buenos Aires
  - Research Site, Caba
  - Research Site, Capital Federal
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Corrientes
  - Research Site, Córdoba
  - Research Site, La Plata
  - Research Site, Rosario
  - Research Site, Santa Fe
- France (6):
  - Research Site, L'Aigle
  - Research Site, Mûrs-Erigné
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Tours
  - Research Site, Vannes
- Germany (12):
  - Research Site, Bad Lauterberg im Harz
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Hamburg
  - Research Site, Heilbronn
  - Research Site, Ludwigshafen
  - Research Site, Mainz
  - Research Site, Pirna
  - Research Site, Schmiedeberg
  - Research Site, Wangen
- Italy (3):
  - Research Site, Perugia
  - Research Site, Pisa
  - Research Site, Roma
- Mexico (4):
  - Research Site, Acapulco
  - Research Site, Guadalajara
  - Research Site, México
  - Research Site, Veracruz
- Netherlands (10):
  - Research Site, Deurne
  - Research Site, Gorinchem
  - Research Site, Groningen
  - Research Site, Lichtenvoorde (gld)
  - Research Site, Losser
  - Research Site, Poortvliet
  - Research Site, Rotterdam
  - Research Site, The Hague
  - Research Site, Wildervank
  - Research Site, Zutphen
- South Africa (7):
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, eMkhomazi
  - Research Site, Johannesburg
  - Research Site, Parow
  - Research Site, Pretoria
  - Research Site, Witbank
- Spain (6):
  - Research Site, Alicante
  - Research Site, Alzira (Valencia)
  - Research Site, Barcelona
  - Research Site, Cornellá de Llobregat (bcn)
  - Research Site, Madrid
  - Research Site, Seville
- Sweden (8):
  - Research Site, Gothenburg
  - Research Site, Järfälla
  - Research Site, Lund
  - Research Site, Malmo
  - Research Site, Skene
  - Research Site, Södertälje
  - Research Site, Stockholm
  - Research Site, Umeå
- United Kingdom (11):
  - Research Site, Addlestone
  - Research Site, Aylesbury
  - Research Site, Bath
  - Research Site, Bolton
  - Research Site, Bury Saint Edmonds
  - Research Site, Cookstown
  - Research Site, Coventry
  - Research Site, Ecclesfield
  - Research Site, Edinburgh
  - Research Site, Mortimer Reading
  - Research Site, Trowbridge

REFERENCES:
- [Result] Nauck MA, Del Prato S, Meier JJ, Duran-Garcia S, Rohwedder K, Elze M, Parikh SJ. Dapagliflozin versus glipizide as add-on therapy in patients with type 2 diabetes who have inadequate glycemic control with metformin: a randomized, 52-week, double-blind, active-controlled noninferiority trial. Diabetes Care. 2011 Sep;34(9):2015-22. doi: 10.2337/dc11-0606. Epub 2011 Aug 4. PMID 21816980
- [Derived] Nauck M, del Prato S, Meier JJ, Duran-Garcia S, Rohwedder K, Elze M, Parikh SJ. [Dapagliflozin versus glipizide as add-on therapy in patients with type 2 diabetes who have inadequate glycemic control with metformin]. Dtsch Med Wochenschr. 2013 Apr;138 Suppl 1:S6-15. doi: 10.1055/s-0032-1305283. Epub 2013 Mar 25. German. PMID 23529570
- See also: CSR-D1690C00004.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=289&filename=CSR-D1690C00004.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The 1st patient was enrolled on 31 Mar 2008. The last patient last visit was on 15 Dec 2009. 1901 patients (pts) were screened and 1217 pts were enrolled with the aim to randomize 816. 2 randomized pts were excluded since they received no medication. Eventually, 814 pts received medication. This study was conducted at 95 centers world-wide.
Pre-assignment Details: For participants with a metformin dose of less than 1500 mg/day, a change in metformin dose in the past 8 weeks or on an Oral Anti-Diabetic (OAD), an 8-week metformin-only dose stabilisation period occurred. A 2-week placebo lead in period occurred after the dose stabilisation period or after enrolment if dose stabilisation period was skipped.
Groups:
- Dapagliflozin Plus Metformin: Experimental dapagliflozin plus metformin
- Glipizide Plus Metformin: Active Comparator glipizide plus metformin
Period: Overall Study
Arm/Group | Dapagliflozin Plus Metformin | Glipizide Plus Metformin
Started | 406 (Of the 406 randomized participants only 400 were included in the full analysis set.) | 408 (Of the 408 randomized participants only 401 were included in the full analysis set.)
Completed | 322 | 314
Not Completed | 84 | 94
Not completed — Incorrect Enrollment | 1 | 1
Not completed — Adverse Event | 33 | 19
Not completed — Subject No Longer Meets Study Criteria | 6 | 27
Not completed — Withdrawal by Subject | 23 | 32
Not completed — Lost to Follow-up | 3 | 3
Not completed — Poor/Non-Compliance | 5 | 1
Not completed — Safety | 1 | 0
Not completed — Death | 1 | 3
Not completed — Various | 11 | 8

BASELINE CHARACTERISTICS:
Population: Full Analysis Set defined as all randomized participants (as randomized) who received at least one dose of double-blind study medication, who have a non-missing baseline value and at least one post-baseline efficacy value for at least one efficacy variable during double-blind treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin Plus Metformin | Glipizide Plus Metformin | Total
Number analyzed (Participants) | 400 | 401 | 801
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (9.37) | 58.6 (9.80) | 58.4 (9.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 179 | 181 | 360
  Male | 221 | 220 | 441
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 27 | 34 | 61
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 24 | 50
  White | 327 | 323 | 650
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 20 | 20 | 40
BMI [Mean (Standard Deviation); unit: kg/m2] | 31.71 (5.104) | 31.23 (5.053) | 31.47 (5.081)
HbA1c [Mean (Standard Deviation); unit: percent] | 7.69 (0.855) | 7.74 (0.886) | 7.72 (0.870)
FPG [Mean (Standard Deviation); unit: ng/mL] | 162.24 (37.796) | 163.91 (41.559) | 163.07 (39.708)

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change in HbA1c Levels
Description: To assess the effect of dapagliflozin plus metformin compared to glipizide plus metformin on the absolute change from baseline in HbA1c level after 52 weeks double-blind treatment in patients with type 2 diabetes who have inadequate glycaemic control on 1500 mg/day or higher doses of metformin therapy alone.
Time Frame: Baseline to Week 52
Population: Full Analysis Set, participants with non-missing baseline and Week 52 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | Dapagliflozin Plus Metformin | Glipizide Plus Metformin
Number analyzed (Participants) | 400 | 401
percent | -0.52 [-0.60 to -0.44] | -0.52 [-0.60 to -0.44]
Statistical Analysis 1: Comparison: Dapagliflozin Plus Metformin vs Glipizide Plus Metformin; The null hypothesis is given as H0: mean(treat) minus mean(reference) >= delta versus the alternative HA: mean(treat) minus mean(reference) < delta (with alpha = 0.025, one-sided); Test type: Non-Inferiority or Equivalence — non-inferior margin delta = 0.35; p < 0.0001, ANCOVA — Significant at alpha=0.025 (1-sided). A hierarchical closed testing procedure was used to control Type I error across the primary & key secondary objectives; with treatment group as effect and baseline value as covariate; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.11 to 0.11], Standard Error of Mean 0.0569

2. Secondary Outcome: Adjusted Mean Change in Body Weight
Description: To assess the effect of dapagliflozin plus metformin compared to glipizide plus metformin on body weight after 52 weeks double-blind treatment.
Time Frame: Baseline to Week 52
Population: Full Analysis Set, participants with non-missing baseline and Week 52 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Dapagliflozin Plus Metformin | Glipizide Plus Metformin
Number analyzed (Participants) | 400 | 401
kg | -3.22 [-3.56 to -2.87] | 1.44 [1.09 to 1.78]
Statistical Analysis 1: Comparison: Dapagliflozin Plus Metformin vs Glipizide Plus Metformin; H0: mean(treat) minus mean(reference) = 0 versus the alternative HA: mean(treat) minus mean(reference) =/= 0; Test type: Superiority or Other; p < 0.0001, ANCOVA — Significant at alpha=0.05 (2-sided). Key secondary endpoints are tested following a hierarchical closed testing procedure; with treatment group as effect and baseline value as covariate; Mean Difference (Final Values) = -4.65, 95% CI 2-sided [-5.14 to -4.17], Standard Error of Mean 0.2483

3. Secondary Outcome: Proportion of Participants With at Least One Episode of Hypoglycemia
Description: To assess the effect of dapagliflozin plus metformin treatment compared to glipizide plus metformin on the occurrence of hypoglycemic events. Least Squares Mean represents the percent of participants adjusted for HbA1c baseline value.
Time Frame: Baseline to Week 52
Population: Full analysis set
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dapagliflozin Plus Metformin | Glipizide Plus Metformin
Number analyzed (Participants) | 400 | 401
Percentage of participants | 3.5 [1.7 to 5.3] | 40.8 [36.1 to 45.5]
Statistical Analysis 1: Comparison: Dapagliflozin Plus Metformin vs Glipizide Plus Metformin; H0: proportion(treat) minus proportion(reference) = 0 versus the alternative HA: proportion(treat) minus proportion(reference) =/= 0; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Based on methodology of Zhang, Tsiatis & Davidian and Davidian, Tsiatis, Zhang & Lu, with adjustment for baseline value; Risk Difference (RD) = -37.2, 95% CI 2-sided [-42.3 to -32.2], Standard Error of Mean 2.578

4. Secondary Outcome: Proportion of Participants With Body Weight Reduction of at Least 5%
Description: To evaluate the effect of dapagliflozin plus metformin compared to glipizide plus metformin on body weight assessed by a reduction after 52 weeks of at least 5% compared to baseline. Least Squares Mean represents the percent of participants adjusted for baseline value.
Time Frame: Baseline to Week 52
Population: Full Analysis Set, participants with non-missing baseline and Week 52 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dapagliflozin Plus Metformin | Glipizide Plus Metformin
Number analyzed (Participants) | 400 | 401
Percentage of participants | 33.3 [28.7 to 37.9] | 2.5 [1.0 to 4.0]
Statistical Analysis 1: Comparison: Dapagliflozin Plus Metformin vs Glipizide Plus Metformin; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Based on methodology of Zhang, Tsiatis & Davidian and Davidian, Tsiatis, Zhang & Lu, with adjustment for baseline value; Risk Difference (RD) = 30.8, 95% CI 2-sided [26.0 to 35.7], Standard Error of Mean 2.480

ADVERSE EVENTS:
Time Frame: Non-serious / serious adverse events on or after the first day and on or prior to the last day of the 52-week double-blind treatment plus 4/30 days or up to follow-up visit if earlier, or up to and including the start date of extension period if earlier.
Description: Participants were questioned at each study visit about the occurrence of any health problems and any examination conducted at a study visit was assessed in comparison to the status at study entry.
Arm/Group | Dapagliflozin Plus Metformin | Glipizide Plus Metformin
Serious Adverse Events (participants affected / at risk) | 35/406 | 46/408
Other Adverse Events (participants affected / at risk) | 163/406 | 260/408
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dapagliflozin Plus Metformin (N=406) | Glipizide Plus Metformin (N=408)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Myocardial Infarction (Cardiac disorders) | 1 | 3
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1
Angina Pectoris (Cardiac disorders) | 1 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Atrioventricular Block Complete (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 1 | 1
Left Ventricular Failure (Cardiac disorders) | 1 | 0
Ventricular Arrhythmia (Cardiac disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Retinal Detachment (Eye disorders) | 1 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Anal Fissure (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Chest Pain (General disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 1
Sudden Death (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic Cirrhosis (Hepatobiliary disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 2
Bronchitis (Infections and infestations) | 1 | 1
Erysipelas (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 1 | 0
Liver Abscess (Infections and infestations) | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Septic Shock (Infections and infestations) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 2
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 1
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 1
Multiple Injuries (Injury, poisoning and procedural complications) | 1 | 0
Postoperative Renal Failure (Injury, poisoning and procedural complications) | 0 | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 1
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 1
Creatinine Renal Clearance Decreased (Investigations) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carotid Artery Stenosis (Nervous system disorders) | 1 | 0
Cerebral Thrombosis (Nervous system disorders) | 1 | 0
Cervicobrachial Syndrome (Nervous system disorders) | 1 | 0
Loss Of Consciousness (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0
Depression Suicidal (Psychiatric disorders) | 0 | 1
Obsessive-Compulsive Disorder (Psychiatric disorders) | 0 | 1
Diabetic Nephropathy (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Urinary Incontinence (Renal and urinary disorders) | 0 | 1
Uterine Prolapse (Reproductive system and breast disorders) | 2 | 0
Alveolitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dapagliflozin Plus Metformin (N=406) | Glipizide Plus Metformin (N=408)
Diarrhoea (Gastrointestinal disorders) | 19 | 26
Nasopharyngitis (Infections and infestations) | 43 | 61
Upper Respiratory Tract Infection (Infections and infestations) | 24 | 31
Influenza (Infections and infestations) | 30 | 30
Urinary Tract Infection (Infections and infestations) | 30 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 21
Dizziness (Nervous system disorders) | 15 | 37
Tremor (Nervous system disorders) | 1 | 31
Headache (Nervous system disorders) | 21 | 17
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 | 27
Hypertension (Vascular disorders) | 30 | 35
Hypoglycemia (Endocrine disorders) | 14 | 162

LIMITATIONS AND CAVEATS:
For participants who did not complete 52 weeks LOCF (last observation carried forward) was used.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an Investigator requests permission to publish data from this study any such publication is to be agreed with AstraZeneca (AZ) in advance. The investigator agrees to provide AZ as soon as possible with drafts of proposed publications. Unless otherwise agreed, AZ shall have a period of 60 days from receipt of the proposed final manuscript to review it and may within such time require that submission for publication of the manuscript be delayed in order for AZ to file patent applications.